CLINICAL TRIAL: NCT04238598
Title: Sham-controlled Randomized Trial of Intra-articular Pulsed Radiofrequency Neuromodulation Versus Intra-articular Steroids for Painful Knee Osteoarthritis
Brief Title: Intra-articular Pulsed Radiofrequency Neuromodulation Versus Intra-articular Steroids for Painful Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center For Interventional Pain and Spine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019IA-PRF
Record Dates: First submitted 2019-10-25; First posted 2020-01-23 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: test, active, control
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active (Active Comparator): intra-articular 4 milliliters 0.5% bupivacaine + 10mg dexamethasone + sham Pulsed Radiofrequency
  Interventions: Procedure: Placebo Intra-Articular Injection
- Control (Placebo Comparator): intra-articular 5 milliliters 0.9% saline + sham Pulsed Radiofrequency
  Interventions: Procedure: Standard of Care Intra- Articular Injection
- Experimental (Experimental): intra-articular 5 milliliters 0.5% bupivacaine + Pulsed Radiofrequency
  Interventions: Procedure: Pulse Radiofrequency

INTERVENTIONS:
Procedure: Pulse Radiofrequency — Two 20-gauge radiofrequency needle with 10mm active tip will be placed intra-articularly from an anterolateral and anteromedial approach to target the medial and lateral compartments. Once satisfactory fluoroscopic placement is noted, the Pulsed Radiofrequency treatment will be administered.
  Arms: Experimental
Procedure: Standard of Care Intra- Articular Injection — Two 20-gauge radiofrequency needle with 10mm active tip will be placed intra-articularly from an anterolateral and anteromedial approach to target the medial and lateral compartments. Once satisfactory fluoroscopic placement is noted, the Intra-Articular treatment will be administered.
  Arms: Control
Procedure: Placebo Intra-Articular Injection — Two 20-gauge radiofrequency needle with 10mm active tip will be placed intra-articularly from an anterolateral and anteromedial approach to target the medial and lateral compartments. Once satisfactory fluoroscopic placement is noted, the Placebo Intra-Articular treatment will be administered.
  Arms: Active

SUMMARY:
To compare the efficacy of intra-articular pulsed radiofrequency to intra-articular steroids in patients with moderate-severe painful osteoarthritis of the knee.

DETAILED DESCRIPTION:
Patients Adult patients with intractable knee pain for more than 6 months and radiographic evidence of grade II, III or IV knee osteoarthritis. Must not have had a knee injection or other interventional procedure for knee pain within the past 12 weeks. Must be on stable medications for the past 12 weeks and willing to keep medications stable for the first 12 weeks of the study.

Study Design Pilot study will enroll 30 patients randomized 1:1:1.

1. Active control - intra-articular 4 milliliters 0.5% bupivacaine + 10mg dexamethasone + sham Pulsed Radiofrequency
2. Placebo control - intra-articular 5 milliliters 0.9% saline + sham Pulsed Radiofrequency
3. Treatment group - intra-articular 5 milliliters 0.5% bupivacaine + Pulsed Radiofrequency

Methods Two 18-gauge radiofrequency needle with 10 millimeter active tip will be placed intra-articularly from an anterolateral and anteromedial approach to target the medial and lateral compartments. Once satisfactory fluoroscopic placement is noted, the Pulsed Radiofrequency or sham-Pulsed Radiofrequency treatment will be administered. Subsequently, the injectate will be administered. Dexamethasone is selected as the corticosteroid as it is colorless and will be indistinguishable from the saline used in the Intra-articular Pulsed Radiofrequency and placebo groups.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving written informed consent
* Patients aged 18 years or older
* Patients with unilateral or bilateral knee pain for at least 3 months
* Radiographic evidence of knee osteoarthritis
* Appropriate candidate for steroid injection as determined by the investigator

Exclusion Criteria:

* Chronic knee pain caused by infection, inflammation, tumors, and fractures
* A history of acute knee pain, previous knee surgery, connective tissue diseases, progressive neurologic disease or uncontrolled psychiatric disorders
* The administration of steroids or hyaluronic acids within the last three months
* Coagulation disorders
* Local infection at the site of intervention planned
* Active litigation related to this pain complaint

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2021-01-19 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analogue Scale pain scores | 1-week, 1-, 3-, 6-, and 12-months
  Evaluates the level of pain. Minimum=0 Maximum=10, Larger number indicates worse outcome

SECONDARY OUTCOMES:
Change in Patient-Reported Outcomes Measurement Information System-29 and Western Ontario and McMaster Universities Osteoarthritis (Index) | 1-week, 1-, 3-, 6-, and 12-months
  Evaluates level of pain. For Patient-Reported Outcomes Measurement Information System-29, Minimum= 8 and Maximum=40. For Western Ontario and McMaster Universities Osteoarthritis (Index), Minimum=0 Maximum=20. Larger number indicates worse outcome
Change in Analgesic use | 1-week, 1-, 3-, 6-, and 12-months
  Evaluates number of medications, doses of medications
Change in Timed Up and Go Test | 1-week, 1-, 3-, 6-, and 12-months
  Evaluates physical mobility
Change in Progression to Surgery | 1-week, 1-, 3-, 6-, and 12-months
  Evaluates effectiveness of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Fishman, MD, Principal Investigator — Center For Interventional Pain and Spine
Locations (1):
- Center for Interventional Pain and Spine, Exton, Pennsylvania, United States